CLINICAL TRIAL: NCT04385641
Title: Study on the Safety and Effectiveness of UCB-NK Cell Infusion in the Treatment of Advanced Gastric Cancer and Gastroesophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Golden Brick Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IH-UCB-NK-422
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: Advanced Gastric Cancer; Gastroesophageal Cancer
Keywords: UCB-NK cell infusion; safety; effectiveness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose-finding (Group A) (Experimental): In this study, the dose was explored according to the "3+3" mode, in which group A was divided into three dose groups: 1.5*10＾9 group, 2*10＾9 group and 3*10＾9 group. If DLT occurs in one of the first three subjects in each dose group within four weeks after cell infusion, three subjects will continue to be included. If more than 1/6 cases of DLT appear in 6 subjects with 1.5*10＾9 dose, the dose level and/or cell infusion frequency and method will be reduced after discussion between the investigator, the collaborator and DMC. If DLT did not occur in the first 3 subjects within 4 weeks after receiving 1.5*10＾9 cell infusion，another three subjects were enrolled into the group received 2*10＾9 cell infusion. DLT did not occur within 4 weeks after cell infusion, it will increase to 3*10＾9 dose group. That is to say, the first three subjects were included for observation for 4 weeks in the 3*10＾9 dose group, if DLT did not occur, there will be another 3 cases, reaching to 6 subjects.
  Interventions: Other: Cell infusion for Dose-finding (Group A)
- Extended research (Group B) (Experimental): If DLT≤1/6, the dose will not be increased. This dose will also be used as the treatment dose of group B. If DLT is more than 1/6 in the 3*10＾9 dose group, three subjects will be added in 2*10＾9 dose group. If DLT ≤1/6 in 4-week observation, the 2*10＾9 will be the maximum tolerable dose, and will be used as the treatment dose of group B. The subjects in group A were enrolled first, after at least 4 weeks of observation for all subjects, six subjects will be included in group B.
  Interventions: Other: Cell infusion for Extended research (Group B)

INTERVENTIONS:
Other: Cell infusion for Dose-finding (Group A) — Group A：HLA-I and HLA-II molecular typing were performed at the serological and molecular levels, and the HLA-I and HLA-II molecular antigens of donor and subjects match on 3, 4, 5 or 6 / 6. After the successful matching, the non myeloablative immunosuppressive pretreatment with cyclophosphamide (900 mg / m＾2 / day) and fludarabine (30 mg / m＾2 / day) will be performed 6, 5, 4 and 3 days before the infusion of UCB-NK cells. After the pretreatment, the cell infusion was started on day 0, and the cell infusion could be divided into 50% and 50% for two consecutive days or every other day. To ensure clinical safety, if treatment-related adverse events reach DLT after the first infusion, the cell infusion will stop.
  Arms: Dose-finding (Group A)
Other: Cell infusion for Extended research (Group B) — Group B：Non myeloablative immunosuppressive pretreatment and cell transfusion were the same as group A.
  Arms: Extended research (Group B)

SUMMARY:
This study is an open, single infusion, cell infusion dose /method exploration study. In patients with gastric cancer and gastroesophageal cancer without effective treatment, the safety of UCB-NK cell immunotherapy was evaluated and the preliminary curative effect results were obtained.

DETAILED DESCRIPTION:
1 Experimental design This study is an open, single infusion, cell infusion dose /method exploration study.

1.1 Screening period (28 days) Screening visit completed within 28 days before the start of the study. The following study process must be completed during screening visits to ensure patient compliance with this study (If the subjects are enrolled, the data collected during the screening period will be taken as the baseline data).

1. Sign informed consent (including consent to provide tumor tissue samples);
2. Record demographic information (including age, nationality, gender);
3. Record past medical history (including smoking history);
4. Record vital signs;
5. Measure height and weight (including BMI);
6. ECOG scores;
7. Physical examination;
8. Gastroscopy examination; 9.12-lead electrocardiogram examination;

10.Cardiac color doppler ultrasound; 11.Laboratory examination (blood routine, blood biochemistry, urine routine, clotting, pregnancy test [women of childbearing age only], infectious diseases); 12.Imaging examination (CT or MRI, enhanced scanning is recommended, MRI is used in patients who are allergic to enhancers); 13.Check inclusion / exclusion criteria; 14.Record adverse events and concomitant medication; 15.Immunogenicity detection; 16.Biomarker detection.

* If these tests have been performed within 28 days prior to the first application, they need not be repeated unless the investigator believes that the patient's tumor load has changed / or the condition requires.

1.2 Pretreatment period (Day - 8 to day - 7)

1. Record vital signs;
2. Measure height and weight (including BMI);
3. ECOG scores.

1.3 Cell infusion stage

1. Record vital signs;
2. Physical examination; 3.12-lead electrocardiogram examination;

4.ECOG scores; 5.Laboratory examination (blood routine, blood biochemistry, urine routine, clotting, pregnancy test [women of childbearing age only], infectious diseases); 6.Imaging examination; 7.Immunogenicity detection; 8.Biomarker detection; 9.Pharmacokinetic blood collection; 10.Administration; 11. Record adverse events and concomitant medication.

1.4 In hospital observation period

1. Record vital signs;
2. Physical examination;
3. Immunogenicity detection;
4. Pharmacokinetic blood collection;
5. Record adverse events and concomitant medication.

1.5 Follow-up (safety and preliminary effectiveness assessment)

After infusion, patients need to return to the hospital for regular examination at the 1st, 2nd, 3rd, 4th, 6th and 12th month (± 7 days), after 12 months, return to hospital for regular inspection every 6 months (±1 month):

1.Record vital signs; 2.Physical examination; 3.12-lead electrocardiogram examination; 4.ECOG scores; 5.Laboratory examination (blood routine, blood biochemistry, urine routine, clotting, pregnancy test [women of childbearing age only], infectious diseases); 6.Imaging examination; 7.Gastroscopy examination (Determine if it is necessary by researchers); 8.Immunogenicity detection; 9.Biomarker detection; 10.Pharmacokinetic blood collection; 11.Record adverse events and concomitant medication.

1.6 Group visit (within 7 days after determination) Regardless of the reasons for the determination of the group, the group visit shall be conducted within 7 days after the determination of the group, and the specific time of the group examination shall be determined by the researcher according to the specific time.

1. Record vital signs;
2. Physical examination; 3.12-lead electrocardiogram examination;

4.ECOG scores; 5.Laboratory examination (blood routine, blood biochemistry, urine routine, clotting, pregnancy test [women of childbearing age only], infectious diseases); 6.Imaging examination; 7.Gastroscopy examination (Determine if it is necessary by researchers); 8.Immunogenicity detection; 9.Biomarker detection; 10.Pharmacokinetic blood collection; 11.Record adverse events and concomitant medication.

2 Research evaluation

2.1 Efficacy endpoint

2.1.1Primary efficacy endpoint

1. Incidence of adverse events during the study period;
2. The incidence of treatment-related adverse events;
3. Incidence of adverse events of special concern;
4. Evaluate DLT.

2.1.2 Secondary efficacy endpoint

1. The peak time, peak value, AUC and survival time of UCB-NK cells after infusion;
2. Objective response rate(ORR);
3. Durative time of remission(DOR);
4. Disease control rate(DCR);
5. Duration of disease control(DDC);
6. Progression free survival(PFS);
7. Overall survival (OS). Other observation index Detection of tumor markers before and after cellular immunotherapy

3 Management of adverse events

3.1 Record

At each visit, all observed or subject mentioned adverse events were accurately recorded by the investigator in the original document and recorded in the "adverse events" page of ECRF. The records include:

1. Name of adverse event;
2. Start date and time;
3. Severity(Level 1, 2, 3, 4, 5);
4. Whether to take measures or not(yes, no)
5. Dose effect on study cell (continuous treatment, temporarily suspended, dose reduction, stop using, end of trial, inappropriate);
6. Relationship with research cell(definitely related, very likely related, possibly related, possibly unrelated, definitely unrelated);
7. Whether it is a serious adverse event or not;
8. Outcome of adverse events(disappearance, remission, persistence, aggravation, death, unknown);
9. Whether the subjects withdraw from the clinical study due to adverse events or not (yes, no).

The researcher shall take corresponding measures according to the adverse events to ensure the safety of the subjects; the institution shall ensure the supply of relevant rescue equipment and drugs to ensure that the corresponding rescue can be given in case of emergency.

4 Statistics

4.1Sample size and calculation basis 18-21 cases of advanced gastric cancer and gastroesophageal cancer is planned to be selected.

Calculation basis: see study design for details.

4.2 Statistical analysis population Full analysis set (FAS): According to the basic principle of intent to analyze (ITT), all subjects who have received at least one trial drug after randomization, excluding those without all data.

Per Protocol Set (PPS): On the basis of FAS set, subjects who met the inclusion and exclusion criteria, completed the administration, and completed the evaluation of main efficacy indicators, had good compliance and did not seriously violate the clinical trial scheme.

Safey Set (SS): All subjects who completed adjuvant chemotherapy after randomization. Safety data will be analyzed based on the actual treatment received.

In this experiment, the baseline data and validity analysis were analyzed by FAS. The main efficacy indicators were analyzed by PP at the same time, giving priority to FAS. Laboratory examination data, adverse events and adverse reactions data were analyzed by SS. The incidence of adverse reactions was calculated with SS as denominator.

5 Test management

5.1 Management and implementation of GCP

1. Both the sponsor and the researcher should implement the quality control and quality assurance system of clinical trials adopting SOP.
2. The original data must meet the requirements of China's GCP.
3. Laboratory test results must be accurate and reliable.
4. All observations and findings should be verified to ensure the reliability of the data.
5. Establish a complete test organization, clear responsibilities of personnel at all levels.
6. The main researchers are responsible for total quality control, perform responsibilities of personnel at all levels.
7. The main researchers are responsible for the design and review of the test scheme and eCRF which are used with the consent of the sponsor and write the summary report after the test.
8. The designated researcher is responsible for formulating the test implementation rules and SOP, which are used in the test.
9. Before the test, the test group will organize all participants to study the program. All participants in the test shall receive GCP training and corresponding certificates.
10. Doctors and nurses participating in the trial should strictly abide by the program, carry out according to the procedure and shall not be changed at will.
11. The designated statistician is responsible for the comprehensive statistical processing of data.

5.2 Supervision system The sponsor will send an inspector to supervise the test together with QA Department of clinical research institution to ensure that the test is carried out in accordance with the scheme and the data recorded in the case record form is the same as the original data. At the same time, the corresponding regulatory agencies may inspect the research center, research database and relevant research documents at their own discretion. The purpose of the audit and inspection is to systematically and independently inspect all research related processes and documents to determine whether the implementation of the clinical study complies with the trial protocol, GCP, declaration of Helsinki and relevant regulatory requirements. The researcher shall inform the sponsor immediately when he receives the inspection notice from the regulatory authority.

5.3 The problems in the research and the countermeasures

1. Revision of the scheme: After the scheme is approved by the ethics committee, a plan of scheme modification shall be prepared in the case of modification, and signed by the main researcher, and the scheme can be modified only with the consent of the sponsor.
2. The scheme with modification can only be implemented after it is reported to the ethics committee, unless it is to solve the security risk faced immediately or only involves logistics and administrative modification.
3. Any personnel participating in the test shall not violate the scheme. In case of any violation of the scheme, a description shall be written and the sponsor shall be informed, the latter has the right to decide whether to continue the test.
4. Any AE or SAE occurred during the test will be declared and handled in accordance with the requirements specified in the program.

5.4 Clinical research data management

1. Researchers must ensure that the data are true, complete and accurate.
2. All items in the research record shall be filled in, and no blank or missing items are allowed. When making any correction, only scribing is allowed, and the modified data shall be noted, give reasons and sign and date by the investigator.
3. Laboratory inspection items should be complete.
4. This test adopts electronic data acquisition (EDC) system for data management, and the name of EDC system is BioKnow-eTMF.
5. Construction of electronic case report form (eCRF): the data manager builds eCRF according to research scheme.
6. EDC system authority control: The sponsor confirms the EDC account list, fills in the account application form and sends it to the data administrator for review, then the data administrator hands over to the database designer to open the account and grant different roles and authorities to the main researchers, researchers, supervisors and auditors to access to EDC.
7. Data entry: eCRF shall be completed by the principal investigator of each center or its authorized research assistant (CRC), CRC needs to input the data in the original record form into eCRF timely and accurately. eCRF is not regarded as the original record, and its content originates from the original record.
8. Logical verification: At the same time of data entry, EDC performs logical verification and issues system query. In addition to the system query, the data administrator manually checks the text data and issues the artificial query if there is a problem.
9. Question and answer: Researchers can answer questions real-time online. The data administrator and the supervisor review the researcher's answers and, if necessary, raise questions again until all questions are resolved.
10. Data lock and export: All patients complete the test and all the original data are input into EDC system. The main researchers, sponsors, statistical analysts and data administrators conduct blind review on data. After confirming that there is no doubt about the data, all parties shall sign the database locking application form, and the data administrator shall lock the database. After locking, the data administrator will export the analysis database to the statistician for statistical analysis. The locked data can no longer be edited. The non key data problems found after the locking can be corrected in the statistical analysis program and the file records can be prepared after confirmation. If there is exact evidence proving that it is necessary to unlock the database, it shall be approved by the sponsor.

5.5 Data record and document retention The data of the subjects on the electronic case report form shall be recorded in code form, and the subjects can only be identified by the number of the subjects or their initials.

All information required by the test scheme must be provided, any omission needs to be justified.

The researcher must keep the original documents of each subject participating in the trial. All information on the electronic case report form must come from these original documents，which should contain all demographic and treatment information, including laboratory test data, ECG, etc., as well as the signed informed consent with test number and subject.

Basic documents must be retained by researchers for the time required by national or international regulations (usually 5 years after the end of clinical study or the final approval of marketing). The sponsor shall inform the research institution of the time when relevant test records are no longer needed.

6 Responsibilities and regulations The sponsor shall provide the researcher with the materials and research funds related to the experiment, such as the researcher's manual, and qualified test drugs and test materials (including: approval documents of drug clinical research, copies of business license, drug production license and GMP certificate of the sponsor, original or copy of drug inspection report). The sponsor and the researcher shall jointly formulate the test scheme, which shall be determined by both parties. According to the test scheme, the researcher conducted the test in accordance with the current national regulations.

The researcher shall keep all information provided by the sponsor strictly confidential, and also require other participants and ethics committee to take the same confidentiality measures. The information provided to the researcher shall not be disclosed to others without the written permission of the sponsor.

All data and results of the test shall be possessed jointly by the researcher and the sponsor. The researcher shall not publish on its own without the consent of the sponsor. Any article to be published shall be submitted to the sponsor before sending out. The sponsor will review its accuracy, confirm that the confidential information has not been disclosed and supplement relevant information.

ELIGIBILITY:
Inclusion Criteria:

* 1)Patients with advanced gastric cancer or gastroesophageal cancer confirmed by pathology and failed in standard treatment; 2)ECOG scores≤1； 3)Expected life>12 weeks； 4)According to RECIST1.1，there is at least one target lesion that can be stably evaluated, defining as: the longest diameter of non lymph node lesions ≥ 10 mm, or the short diameter of lymph node ≥ 15mm; 5)Sufficient vein access for monocyte collection; 6)Hematology parameters meet the following requirements: Neutrophil absolute value≥1.5×109 / L; Leukocyte≥4.0×109 / L; Hemoglobin≥80g / L; Platelets≥75×109 / L; 7) Liver function meets the following conditions: Total bilirubin≤1.5×ULN (no liver metastasis); Aspartate aminotransferase≤2.5×ULN (no liver metastasis); Alanine aminotransferase≤2.5×ULN (no liver metastasis); Alkaline phosphatase≤2.5×ULN (no liver metastasis); Total bilirubin≤2×ULN (with liver metastasis); Aspartate aminotransferase≤5.0×ULN (with liver metastasis); Alanine aminotransferase≤5.0×ULN (with liver metastasis); Alkaline phosphatase≤5.0×ULN (with liver metastasis); 8) Renal function meets the following conditions: Serum creatinine≤1.5×ULN; 9) Coagulation function meets the following conditions: International standardization ratio (INR) ≤1.5; Apart prothrombin (PTT或 APTT) ≤1.5×ULN; 10) Heart function meets the following conditions: Left ventricular ejection fraction (LVEF)≥50%; 11) The subjects can communicate well with the researchers and follow the visit, treatment, laboratory examination and other relevant regulations; 12) Female and male subjects of childbearing age agree to take effective contraceptive measures throughout the study period up to 6 months after completion of administration; 13) The subjects must give informed consent to the study before the trial and sign the written informed consent voluntarily.

Exclusion Criteria:

* 1)Serious or uncontrollable heart disease,including: Congestive heart failure with NYHA grade 3 or 4； Unstable angina beyond the control of drugs； History of myocardial infarction six months before the selection; Serious arrhythmia requiring medication; 2)Other malignant tumors occurred in the past 5 years; 3)≥ grade 3 peripheral neuropathy; 4)Patients with active infections (viruses, bacteria or fungi) requiring special treatment 5) Active hepatitis B or hepatitis C; current or past alcoholism; cirrhosis; 6)Human immunodeficiency virus ( HIV) positive; 7)According to the judgment of researchers, uncontrollable systemic diseases, including: diabetes, hypertension, pulmonary fibrosis, acute lung disease, interstitial lung disease, glaucoma, immune disease, pleural effusion or peritoneal effusion with symptoms requiring drainage, etc; 8)Pregnant or lactating women; 9)Baseline measurement, QTc interval, male > 450 ms, female > 470 ms; 10)Other unsuitable conditions judged by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-10-08 (Estimated); Study Completion 2022-10-08 (Estimated)

PRIMARY OUTCOMES:
Safety assessment | 4 weeks
  Evaluation of adverse events and severity according to CTCAE v5.0
Hematology toxicity | 7 days
  After 7 days of treatment, the ≥ 4 degree hematotoxicity (excluding lymphocyte reduction) related to UCB-NK treatment could not recover to ≤ 3 degree
Non hematologic toxicity | 7 days
  Any non hematologic toxic reaction≥4 degree related to UCB-NK treatment cannot be reduced to≤3 degree within 3 days and no further improvement is found; Gastric mucosal injury including gastric hemorrhage≥3 degree related to UCB-NK treatment; Other non hematologic toxicity≥3 degree related to UCB-NK treatment lasted for more than 7 days.

SECONDARY OUTCOMES:
Tumor assessment | 4 years
  Imaging of the chest, abdomen and pelvis (either enhanced CT or MRI) and tumor markers should be obtained at baseline (before the pretreatment of first lymphocyte clearance)， this imaging evaluation is the baseline examination of this study. After the infusion, patients need to return to the hospital at the 1st, 2nd, 3rd, 4th, 6th and 12th month (± 7 days) and every 6 months (± 1 month) after the 12th month to check the imaging of chest, abdomen and pelvis and tumor markers. Follow up to the disease progress, unwilling to be followed up, loss of follow-up, death or the end of the study, whichever occurs first.
  Imaging evaluation is up to the established disease progression (PD) according to the RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Changguo hospital of Zibo, Zibo, China